CLINICAL TRIAL: NCT03799263
Title: A Six Minute Walking Test Based Index as an Outcome Predictor in COPD Subjects
Brief Title: A Six Minute Walking Test Based Index as an Outcome Predictor in COPD Subjects. (Chronic Obstructive Pulmonary Disease)
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maugeri Foundation (Other)
Collaborators: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, elisabetta zampogna, Dr, Maugeri Foundation
Other Study IDs: 2019001
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: COPD; Mortality; Disease Exacerbation; Exercise Capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: evaluation group — Recordings Pneumologic assessment Severity grades (I-IV: old GOLD and A-D: new GOLD) Smoke History Drug therapy Comorbidities 6MWT performed within previous 10-14 months, if available. Measurements Standard exams usually performed at Rehab Center Lung Function tests and diffusing capacity of the lung for carbon monoxide Arterial Blood Gases Dyspnoea Health Status and Health Related Quality of Life Daily activity Lower limb muscle strength Exercise capacity

SUMMARY:
The six minute walking test (6MWT) is a recognized clinical test to evaluate exercise capacity in different diseases and different conditions. The modalities of performance are described in International Guidelines. The usually reported measure is the distance in meters walked in 6 minutes. Despite the report of a single variable during the test is considered as a limit, changes in monitored variables are seldom analyzed together with the distance walked. In the past there have been some attempts of multifactorial evaluation of 6MWT, however up to date, there is no system considering together the changes of different variables. The investigators wonder whether a multidimensional index based on variables monitored during the 6MWT would better predict 24 month exacerbations and mortality in COPD patients.

DETAILED DESCRIPTION:
Rationale: the six minute walking test (6MWT) is a recognized clinical test to evaluate exercise capacity in different diseases and different conditions. In COPD patients the 6MWT is a marker of severity, influenced by the severity of airway obstruction as well as of comorbidities. This test has been shown as a predictor of survival and need of hospitalization. The modalities of performance are described in International Guidelines. The usually reported measure is the distance in meters walked in 6 minutes. However, besides the pathological conditions, this result is influenced by the individual demographic and anthropometrics characteristics. The Minimal Clinically Important Difference in COPD subjects is reported to be 30 meters (m.). A decrease greater than 30 m., as compared to the previous year, is a predictor of death risk. During the test some physiological variables should be monitored such as heart rate (HR), and pulse oxymetry (SpO2). An oxyhemoglobin desaturation >4% or a SpO2 <90% during the test, are also predictors of increased risk of death or hospitalization. In addition, also the difference between the HR at baseline and that after one minute after the end of the test (recovery heart rate: HRR) seems to be a predictor of survival and COPD exacerbation rates. Despite the report of a single variable during the test is considered as a limit, changes in monitored variables are seldom analyzed together with the distance walked. In the past there have been some attempts of multifactorial evaluation of 6MWT, however up to date, there is no system considering together the changes of different variables. We wonder whether a multidimensional index based on variables monitored during the 6MWT would better predict 24 month exacerbations and mortality in COPD patients.

Objectives:

Primary Objective: To develop and validate a multidimensional index in COPD subjects with different grades of severity as assessed by the Global Initiative for Chronic Obstructive Lung disease as a predictor of 24 month exacerbation rate.

Secondary Objectives: To evaluate the predictive value of 24 month mortality. To evaluate the relationship of this index and other accepted clinical predictors.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis and grades of severity as assessed by the "old" (I to IV) and "new" (A to D) GOLD guidelines (23)
* Under inhaler therapy for ≥30 days according to guidelines (23)
* Smokers or o ex-smokers, smoke history ≥10 pack/years (p/y)
* Informed Consent Signature.

Exclusion Criteria:

* Associated Comorbidities with short term severe prognosis
* Actual Cardiac Arrythmias
* Pace-maker
* Other associated respiratory diseases
* Chronic Heart Failure New York Heart Association classes III, IV.
* Use of drugs influencing the heart rate
* Changes in drug therapy in the previous 30 days
* Use of systemic steroids or antibiotics in the previous 30 days
* Unscheduled visits or admission to the Emergency Room for symptoms worsening in the previous 30 days
* Pneumonia during the previous 60 days
* Myocardial Infarction in the previous 4 months
* Subjective and objective inability to perform the 6MWT
* Inability to carry the oxygen cylinder.

Ages: 45 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stable COPD patients assessed for Pulmonary Rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
COPD Exacerbation | 24 month
  number of patients with acute exacerbations (treated with antibiotics or steroids)
Mortality | 24 month
  number of patients died

SECONDARY OUTCOMES:
hospitalizations | 24 month
  number of patients hospitalized for COPD
symptoms and anthropometrics characteristics correlation | 24 month
  Index correlation capacity with dyspnoea (Medical Research Council questionnaire, Barthel Dyspnoea), body weight (kilogram), heart frequency (HR), distance walked (6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, Prof, Study Director — Maugeri Foundation
Locations (1):
- Maugeri Foundation, Tradate, VA, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Butland RJ, Pang J, Gross ER, Woodcock AA, Geddes DM. Two-, six-, and 12-minute walking tests in respiratory disease. Br Med J (Clin Res Ed). 1982 May 29;284(6329):1607-8. doi: 10.1136/bmj.284.6329.1607. No abstract available. PMID 6805625
- [Result] Spruit MA, Watkins ML, Edwards LD, Vestbo J, Calverley PM, Pinto-Plata V, Celli BR, Tal-Singer R, Wouters EF; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) study investigators. Determinants of poor 6-min walking distance in patients with COPD: the ECLIPSE cohort. Respir Med. 2010 Jun;104(6):849-57. doi: 10.1016/j.rmed.2009.12.007. Epub 2010 May 14. PMID 20471236
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Lama VN, Flaherty KR, Toews GB, Colby TV, Travis WD, Long Q, Murray S, Kazerooni EA, Gross BH, Lynch JP 3rd, Martinez FJ. Prognostic value of desaturation during a 6-minute walk test in idiopathic interstitial pneumonia. Am J Respir Crit Care Med. 2003 Nov 1;168(9):1084-90. doi: 10.1164/rccm.200302-219OC. Epub 2003 Aug 13. PMID 12917227
- [Result] Rodriguez DA, Kortianou EA, Alison JA, Casas A, Giavedoni S, Barberan-Garcia A, Arbillaga A, Vilaro J, Gimeno-Santos E, Vogiatzis I, Rabinovich R, Roca J. Heart Rate Recovery After 6-min Walking Test Predicts Acute Exacerbation in COPD. Lung. 2017 Aug;195(4):463-467. doi: 10.1007/s00408-017-0027-0. Epub 2017 Jun 17. PMID 28624883
- [Result] Puhan MA, Mador MJ, Held U, Goldstein R, Guyatt GH, Schunemann HJ. Interpretation of treatment changes in 6-minute walk distance in patients with COPD. Eur Respir J. 2008 Sep;32(3):637-43. doi: 10.1183/09031936.00140507. Epub 2008 Jun 11. PMID 18550610